CLINICAL TRIAL: NCT02731950
Title: The Analgesic Efficacy of Magnesium Sulfate as an Adjuvant to Continuous Presternal Bupivacaine Infusion Through a Single Catheter After Cardiac Surgery; A Prospective Randomized Double Blind Study.
Brief Title: Presternal Bupivacaine Plus Magnesium Sulfate Infusion After Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Lecturer of Anesthesia and critical care Medicine, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB00009904
Record Dates: First submitted 2016-03-26; First posted 2016-04-08 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Pain; Postoperative Pain
Keywords: Sternotomy , cardiac surgery , pain
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A magnesium (Active Comparator): Consists of 20 patients:
  Each receive bupivacaine 0.125% with 5% magnesium sulfate by infusion through a small diameter multi-hole soft catheter generally used for epidural analgesia positioned anterior to the sternum above the fascia in the subcutaneous tissue during wound closure for 48 hours postoperative. A bolus of 5 ml of the study solution will be injected in the catheter after aspiration test before connection to infusion pump that delivers continuous infusion pump that delivers continuous infusion at a fixed rate of 5 ml/h.
  postoperative : 25 µg fentanyl for breakthrough pain. placebo will be given in same intravenous instead of paracetamol and ketorolac of group B , to keep the investigator blinded
  Interventions: Drug: Magnesium Sulfate and Bupivacaine 0.125%
- B control (No Intervention): Consists of 20 patients:
  saline as placebo infusion through a small diameter multi-hole soft catheter positioned anterior to the sternum above the fascia in the subcutaneous tissue during wound closure for 48 Postoperative pain control will be managed with 1gm paracetamol /6 hr, Ketorolac 30 mg every 8-12 hour .25 µg fentanyl for breakthrough pain.

INTERVENTIONS:
Drug: Magnesium Sulfate and Bupivacaine 0.125% — Each patient will receive bupivacaine 0.125% with 5% magnesium sulphate by infusion through a catheter used for epidural analgesia, positioned presternal.
  Other Names: study
  Arms: A magnesium

SUMMARY:
Effective pain relief after cardiac surgery has assumed importance with the introduction of fast track discharge protocols that requires early weaning from mechanical ventilation. Inadequate pain control reduces the capacity to cough, mobility, increases the frequency of atelectasis, and prolongs recovery. Infiltration of local anesthetics near the surgical wound has shown to improve early postoperative pain in various surgical procedures.

Magnesium is the fourth most plentiful cation in our body. It has antinociceptive effects in animal and human models of pain.

DETAILED DESCRIPTION:
Effective pain relief after cardiac surgery has assumed importance with the introduction of fast track discharge protocols that requires early weaning from mechanical ventilation. Inadequate pain control reduces the capacity to cough, mobility, increases the frequency of atelectasis, and prolongs recovery.

A major cause of pain after cardiac surgery is the median sternotomy particularly on the first two postoperative days.

The most often used analgesics in these patients are parenteral opioids which can lead to undesirable side-effects as sedation, respiratory depression, nausea, and vomiting.

Infiltration of local anesthetics near the surgical wound has shown to improve early postoperative pain in various surgical procedures.

Magnesium is the fourth most plentiful cation in our body. It has antinociceptive effects in animal and human models of pain.

It has been mentioned in a systematic review that it may be worthwhile to further study the role of supplemental magnesium in providing perioperative analgesia, because this is a relatively harmless molecule, is not expensive and also because the biological basis for its potential antinociceptive effect is promising.

These effects are primarily based on physiological calcium antagonism, that is voltage-dependent regulation of calcium influx into the cell, and noncompetitive antagonism of N-methyl-D-aspartate (NMDA) receptors.

postoperative pain control will be by 1gm paracetamol / 6 hr, Ketorolac tromethamine 30 mg / 8:12 hour in control group vs bupivacaine 0.125% plus magnesium sulfate 5% through a single catheter after parasternal block in in study group after cardiac surgery.

The investigators primary outcome is pain scores assessment , the secondary outcomes are extubation time, postoperative respiratory parameters, serum cortisol level

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* American Society of Anesthesiologists physical status II and III
* Patients scheduled for open heart surgery with sternotomy

Exclusion Criteria:

* Emergency surgery
* Clinically significant kidney or liver disease
* Patients allergic to local anesthetic
* Patients with prolonged CPB time (>120 min)
* Patients required intra-aortic balloon pump

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment using a VAS | up to day 2 postoperative
  Pain score postoperatively on patient's arrival at the ICU, every 4 h for 12 h then every 6 h for 48 h using a VAS (0 = no pain, 10-the worst pain imaginable)

SECONDARY OUTCOMES:
serum cortisol level | first and second postoperative day
  assessing evening serum cortisol

CONTACTS AND LOCATIONS:
Overall Officials: Emad Zarief Kamel Said, MD, Study Director — Assiut University
Locations (1):
- Emad Zarief Kamel Said, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided